CLINICAL TRIAL: NCT06803550
Title: Effect of Enhanced Recovery After Surgery in Reducing the Incidence of Postoperative Urinary Retention After Surgery for Benign Anorectal Conditions: a Randomized Controlled Trial
Brief Title: Effect of Enhanced Recovery After Surgery for Benign Anorectal Conditions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mostafa shalaby, MD, MSc, PhD, Associate Professor & Consultant Colorectal Surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R.24.11.2877
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Anal Fistula; Anal Fissure Chronic; Haemorrhoid; Enhanced Recovery After Surgery (ERAS) Protocol
Keywords: ERAS; Postoperative urinary retention; Benign anorectal conditions; Anal fistula; Anal fissure; Haemorrhoids
MeSH Terms: conditions — Rectal Fistula; Hemorrhoids; Fissure in Ano

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced recovery after surgery protocol (Active Comparator): ERAS pathway was developed based on the available guidelines and protocols it includes 14 items
  Interventions: Other: Enhanced recovery after surgery protocol
- Routine practice (Other): This is the routine preoperative preparation
  Interventions: Other: Routine pathway

INTERVENTIONS:
Other: Enhanced recovery after surgery protocol — ERAS pathway was developed based on the available guidelines and protocols it includes 14 items:
  1. Preoperative patient education using an information sheet which includes instructions on postoperative wound care, pain management, and preventing and managing constipation.
  2. Single preoperative enema 2 hours prior to surgery.
  3. Solid or semisolid food stopped 6 hours before surgery.
  4. Clear liquids may be continued up to 2 hours before surgery.
  5. Preoperative carbohydrate loading in non-diabetic patients for up to 2 hours prior to surgery in the form of a single 330 ml high-carbohydrate clear drink (apple juice).
  6. Saddle anesthesia.
  7. Single dose of intravenous 500 mg metronidazole at the time of the anaesthesi induction.
  8. Restriction of intraoperative intravenous fluids to less than 500 ml.
  9. Balanced chloride-restricted crystalloid solutions should be used for maintenance infusions and fluid boluses.
  10. A bundle measures to reduce surgical site infection which includes
  Arms: Enhanced recovery after surgery protocol
Other: Routine pathway — This is the routine preoperative preparation at our institute
  Arms: Routine practice

SUMMARY:
This study aims to assess the role of Enhanced recovery after surgery(ERAS) protocol in reducing postoperative urine retention (POUR) after surgery for benign anorectal conditions.

DETAILED DESCRIPTION:
This study aims to assess the role of Enhanced recovery after surgery(ERAS) protocol in reducing postoperative urine retention (POUR) after surgery for benign anorectal conditions.

Patients of both sexes aged between 18 and 90 years old presented; with benign anorectal conditions including chronic anal fissure, hemorrhoids, and fistula-in-ano will be eligible for the study.

Eligible patients will be randomized in equal proportions to RRAS or ROUTINE pathways. The ERAS pathway was developed based on the available guidelines and protocols it includes 14 items.

Patients allocated to ERAS pathway must fulfill all the 14 items. The ROUTINE pathway will represent the routine practice which may include certain ERAS items or those who will not fulfill the 14 items.

For the end points of the study, all patients will be followed-up by a phone call 72 hours postoperatively then in the outpatients' department for a period of a total of 30 days postoperatively. However, patients will be advised to visit the outpatients' department at any other time during the trial if they developed any unfavorable event.

The primary outcome will be the 72-hours postoperative urinary retention after anorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* both sexes
* aged between 18 and 65 years old
* presented with benign anorectal conditions including chronic anal fissure, hemorrhoids, and fistula-in-ano will be eligible for the study

Exclusion Criteria:

* younger than 18
* older than 65 years old
* pregnant female
* history of relevant urological diagnosis (benign prostatic hyperplasia/prostate cancer/urethral stricture/bladder neck stenosis/detrusor underactivity/detrusor overactivity)
* history of relevant urological procedure (radical prostatectomy/ transurethral prostatectomy/bladder neck or urethral surgery/pelvic radiotherapy)
* use of permanent urinary catheter
* intraoperative urological procedures
* with any form of urinary diversion
* severe cognitive impairment
* who undergo other anorectal procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
72-hours postoperative urinary retention after anorectal surgery | 72 hours after surgery
  the inability to void, with the patient needing bladder decompression by catheterization as determined by the treating clinician within 1 week of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Shalaby, MD, PhD, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University Hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No